CLINICAL TRIAL: NCT01629446
Title: A Single-Center, Open-Label, Single-Period, Single-Treatment Study to Determine the Mass Balance of a Single Oral Dose of 14C Labeled Lofexidine
Brief Title: Lofexidine Mass Balance in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: USWM, LLC (dba US WorldMeds) (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: USWM-LX1-1003-1; 1R01DA030916-01 (Other Grant/Funding Number: National Institute on Drug Abuse)
Record Dates: First submitted 2012-06-14; First posted 2012-06-27 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Normal Healthy Volunteers
Keywords: Phase 1; Normal healthy volunteers; Mass Balance
MeSH Terms: interventions — lofexidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lofexidine HCl with 14C tracer (Experimental)
  Interventions: Drug: Lofexidine hydrochloride

INTERVENTIONS:
Drug: Lofexidine hydrochloride — Single Dose = Solution containing 400 μg lofexidine HCl and a tracer amount of 14C lofexidine

SUMMARY:
The purpose of this study is to see how lofexidine (investigational study formulation drug) is absorbed, broken down, and removed from the body. To do this, a special form of the study drug will be used that has a radioactive carbon atom attached. Blood, urine, and feces samples will be collected at different times to measure the amount of the study drug and radioactivity they contain. The amount of radioactivity you will be exposed to is less than the amount of radiation from a regular X-ray.

DETAILED DESCRIPTION:
The purpose of this study is to determine the mass balance of a single oral dose of 14C labeled lofexidine. Study US WorldMeds Reference Number USWM-LX1-1003, conducted in July and August of 2011, was a single-center, open-label, two-period, two-treatment, randomized sequence study to determine the mass balance and absolute bioavailability of a single oral dose of 14C-labeled lofexidine compared to a single intravenous dose of lofexidine. During the conduct of the study, deficiencies occurred in the collection and processing of urine samples from subjects administered the oral dose of 14C-labeled lofexidine. In study USWM-LX1-1003-1, six male subjects will be dosed with 14C labeled lofexidine oral solution in order to provide accurate data for the mass balance portion of the study. Male subjects who successfully participated in and completed study USWM-LX1-1003 will be enrolled first. Additional male subjects will be enrolled as needed to provide a cohort of 6 subjects. Additional provisions to ensure adequate urine collections have now been implemented at the site and will be utilized in USWM-LX1-1003-1. All blood draws for pharmacokinetic analysis and radioanalysis, and all urine and fecal collection intervals, will occur at the same time points in USWM-LX1-1003-1 as they did in USWM-LX1-1003.

To study the absorption, distribution, metabolism, and elimination (ADME), trace amounts of 14C compounds are quantified using accelerator mass spectrometry (AMS). As a form of an isotope ratio atom counter that achieves the lowest detection limits of any type of mass spectrometry, AMS provides quantitative sensitivity towards 14C labeled compounds to low attomole (10-18) levels. This high degree of sensitivity enables the detection of compounds in very small specimens and/or tissues after administration of doses that can be both chemically and radiochemically small (microdose levels).

At the radioactive dose to be given (approximately 280 nCi; 10.36 kBq) the total radiation exposure to the participant is within the level of background radiation exposure that occurs naturally and orders of magnitude (1000 fold reduction on average) below the levels typical for human metabolism studies using 14C tracers.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a male
* Subject must be between 18 and 50 years of age (inclusive).
* Subject's Body Mass Index (BMI) must be between 18 and 30 kg/m2 (inclusive), and subject must weigh a minimum of 50 kg (110 lbs).
* Subject must voluntarily consent to participate in this study and provide their written informed consent prior to start of any study-specific procedures.
* Subject is willing and able to remain in the study unit for the entire duration of each confinement period.
* Subject's vital signs must be within the following ranges to be included: Vital signs measured sitting after 3 minutes rest; heart rate: 50-90 bpm; systolic BP: 100-140 mmHg; and diastolic BP: 50-90 mmHg. Out-of-range vital signs may be repeated once. Predose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) prior to study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval prior to dosing.
* Subject is willing to eat entire meals and snacks provided during confinement at the research facility; and understand that the diet will include foods with high fiber content and possibly prune juice.
* Subject is willing to remain in the clinical research center for a minimum of 7 consecutive days during pre-dose, dose, and post-dose evaluation periods.
* Subject is willing to collect all urine and fecal samples for the duration of the study period as required.
* Subject is willing to use a waterless commode located in a designated dry room for urine and feces collection for the duration of the study period as required.
* Subject is willing to abstain from showering for the first 72 to 96 hours following dose administration. After the restriction from showering is lifted, subject must be willing to provide a urine sample prior to showering for the remainder of the confinement period.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* Has a clinically significant abnormal finding on the physical exam, medical history, ECG, or clinical laboratory results at screening.
* History of any syncopal episode or seizures.
* Presence of acute disease state (eg, nausea, vomiting, fever, diarrhea) within 7 days prior to scheduled dose administration.
* History or presence of allergic or adverse response to lofexidine or related drugs.
* Has been on a significantly abnormal diet during the 4 weeks preceding the first dose of study medication.
* Has donated blood or plasma within 30 days prior to the first dose of study medication.
* Has participated in a standard radiolabeled clinical trial within the last 12 months prior to the first dose of study medication or a micro tracer clinical trial within the last 3 months prior to the first dose of study medication.
* Has participated in another clinical trial (randomized subjects only) within 30 days prior to the first dose of study medication.
* Has used any over-the-counter (OTC) medication, including nutritional supplements, within 7 days prior to the first dose of study medication.
* Has used any prescription medication within 14 days prior to the first dose of study medication.
* Has been treated with any known drugs that are moderate or strong inhibitors/inducers of CYP enzymes such as barbiturates, phenothiazines, cimetidine, carbamazepine, etc., within 30 days prior to the first dose of study medication and that in the Investigator's judgment may impact subject safety or the validity of the study results.
* Has smoked or used tobacco products within 60 days prior to the first dose of study medication.
* Has any prior history of substance abuse or treatment (including alcohol) within the past 2 years.
* Has a positive urine screen for drugs of abuse (amphetamines, barbiturates, benzodiazepines, cocaine, cannabinoids, opiates).
* Has had a positive test for, or has been treated for hepatitis B, hepatitis C, or Human Immunodeficiency Virus (HIV).
* Has orthostatic hypotension at screening defined as a drop in systolic blood pressure ≥ 20 mmHg or a fall in diastolic blood pressure ≥ 10 mmHg following a 2 minute stand. Out-of-range vital signs may be repeated once. Predose vital signs will be assessed by the Principal Investigator or designee (e.g., a medically qualified sub-investigator) prior to study drug administration. The Principal Investigator or designee will verify the eligibility of each subject with out-of-range vital signs and document approval prior to dosing.
* Subjects with a QTcF greater than 450 msec at screening obtained after 5 minutes rest in a supine position using the ECG machine algorithm. The ECGs may be repeated as appropriate in order to confirm values and rule out extraneous results.
* Has irregular bowel habits. ("Irregular" being defined for the purpose of this study as NOT having a bowel movement at least every 2 days.)
* Has been exposed to radiation, including dental or medical imaging such as x ray or tomography, in the 6 months prior to dose administration.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Mass Balance | plasma, urine, and fecal samples up to 216 hours post dose
  To study the absorption, distribution, metabolism, and elimination (ADME), trace amounts of 14C compounds are quantified using accelerator mass spectrometry (AMS). As a form of an isotope ratio atom counter that achieves the lowest detection limits of any type of mass spectrometry, AMS provides quantitative sensitivity towards 14C labeled compounds to low attomole (10-18) levels. This high degree of sensitivity enables the detection of compounds in very small specimens and/or tissues after administration of doses that can be both chemically and radiochemically small (microdose levels).

SECONDARY OUTCOMES:
tolerability of lofexidine oral solution | plasma samples over 144 hours post dose
  To determine the tolerability of lofexidine oral solution, plasma samples will be collected over 144s period post dose. Plasma samples will be collected for possibly pharmacokinetic analysis; radioanalysis samples will be analyzed for combined lofexidine and metabolites using a validated analytical method.

CONTACTS AND LOCATIONS:
Overall Officials: James A Longstreth, PhD, Principal Investigator — US WorldMeds; Charles W Gorodetzky, MD, PhD, Principal Investigator — US WorldMeds; Mark Leibowitz, MD, Principal Investigator — Worldwide Clinical Trials
Locations (1):
- Worldwide Clinical Trials, San Antonio, Texas, United States